CLINICAL TRIAL: NCT00184353
Title: In Vivo Proton MR Spectroscopy of Brain Metastases Obtained at 1,5T and 3T.
Brief Title: Clinical MR Spectroscopy of Brain Metastases at 1,5T and 3T.
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: 173-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Neoplasm Metastases
Keywords: brain metastasis; signal to noise ratio; spectral resolution
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- brain metastases: 6 patients
- healthy: 13 volunteers

SUMMARY:
Increasing magnetic field is known to give improvements in signal-to-noise-ratio (SNR) and spectral resolution. To investigate this, spectra from different subjects were examined using two clinical MR instruments operating at 1.5T and 3T respectively.

ELIGIBILITY:
Inclusion Criteria:

* brain metastases

Exclusion Criteria:

* children
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastases
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2003-11; Primary Completion 2004-12 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Lundgren, MD PhD, Study Director — Cancer Clinic, St.Olavs Hospital Trondheim University Hospital; Ingrid S Gribbestad, PhD, Study Chair — Norwegian University of Science and Technology, Faculty of Medicine
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Sjobakk TE, Lundgren S, Kristoffersen A, Singstad T, Svarliaunet AJ, Sonnewald U, Gribbestad IS. Clinical 1H magnetic resonance spectroscopy of brain metastases at 1.5T and 3T. Acta Radiol. 2006 Jun;47(5):501-8. doi: 10.1080/02841850600644808. PMID 16796315